CLINICAL TRIAL: NCT06712615
Title: A Phase II Randomized, Double-blind, Multi-center Study to Investigate the Efficacy and Safety of PG-102(MG12) Compared With Placebo in Subjects With Obesity and in Subjects With Type 2 Diabetes Mellitus (T2DM)
Brief Title: Phase II Study of PG-102(MG12) Compared With Placebo in Obesity and Type 2 Diabetes
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ProGen. Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PG-102-P2-01
Record Dates: First submitted 2024-11-26; First posted 2024-12-02 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Type 2 Diabetes Mellitus (T2DM); Obesity Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Investigator)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Cohort A (Experimental): Cohort A will include two sub-cohorts with different dosing schedules in participants diagnosed with type 2 diabetes.
  Interventions: Biological: PG-102
- Cohort B1 (Experimental): Cohort B1 will include two sub-cohorts with different dosing schedules in participants with obesity.
  Interventions: Biological: PG-102
- Cohort B2 (Experimental): Cohort B2 will include two sub-cohorts with different dosing schedules in participants with obesity and type 2 diabetes.
  Interventions: Biological: PG-102
- Cohort A (Placebo) (Placebo Comparator): Cohort A will include two sub-cohorts with different dosing schedules in participants diagnosed with type 2 diabetes.
  Interventions: Other: Placebo
- Cohort B1 (Placebo) (Placebo Comparator): Cohort B1 will include two sub-cohorts with different dosing schedules in participants with obesity.
  Interventions: Other: Placebo
- Cohort B2 (Placebo) (Placebo Comparator): Cohort B2 will include two sub-cohorts with different dosing schedules in participants with obesity and type 2 diabetes.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: PG-102 — * Participants will receive PG-102 by subcutaneous (SC) injection.
  * Other Names: MG12
  Arms: Cohort A; Cohort B1; Cohort B2
Other: Placebo — Participants will receive placebo by SC injection
  Arms: Cohort A (Placebo); Cohort B1 (Placebo); Cohort B2 (Placebo)

SUMMARY:
This is a Phase 2, therapeutic exploratory study designed to evaluate the safety and efficacy of PG-102 compared with placebo. Part A includes Cohort A, comprising participants with type 2 diabetes mellitus (T2DM). Part B includes two cohorts: Cohort B1, enrolling participants with obesity, and Cohort B2, enrolling participants with both obesity and T2DM.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 19 to 75 years who provide informed consent.

   [Part A: Type 2 Diabetes Mellitus (T2DM) Specific Criteria]
2. Diagnosed with type 2 diabetes for at least 6 months, with HbA1c between 7.0% and 10.0%, despite adherence to diet and exercise therapy according to diabetes treatment guidelines.
3. Stable on metformin monotherapy or metformin in combination with one oral hypoglycemic agent for at least 90 days.
4. BMI between 18.5 kg/m² and 30.0 kg/m², with a minimum weight of 55 kg for men and 50 kg for women.

   [Part B: Obesity (OB) Specific Criteria]
5. Failed at least one attempt at weight loss through diet and exercise.
6. Cohort B1: BMI ≥ 30 kg/m²
7. Cohort B2: BMI ≥ 27 kg/m² 8-1. Cohort B2: Diagnosed with type 2 diabetes for at least 6 months, with HbA1c between 7.0% and 10.0%.

8-2. Cohort B2: Received treatment with diet and exercise alone, OR stable on approved oral antidiabetic monotherapy or combination therapy for at least 90 days prior to screening.

Exclusion Criteria:

1. Participation in another clinical trial within 90 days.
2. Known hypersensitivity to study drugs or their components.
3. Inability to administer the drug in the abdomen.
4. History of severe gastrointestinal disorders, recent obesity-related surgeries, or conditions affecting gastric emptying.
5. Uncontrolled severe hypertension, hypertriglyceridemia, or severe cardiovascular disease.
6. History of acute pancreatitis, recent cancer, or endocrine disorders causing obesity.
7. Abnormal lab results, including eGFR < 60 mL/min/1.73 m², AST/ALT > 3x ULN, or abnormal ECG.
8. Substance abuse or significant psychiatric disorders within the last 2 years.
9. Pregnant, breastfeeding, or unwilling to use contraception during the study.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Change in Glycated Hemoglobin (HbA1c) in Cohort A | Baseline at weeks 14
Percent Change from Baseline in Body Weight in Cohort B1 and B2 | Baseline at weeks 14

SECONDARY OUTCOMES:
Incidence of Treatment-emergent adverse events (TEAEs) in Cohort A and Cohort B1, B2 | Baseline to weeks 20
Change from Baseline in HbA1c in Cohort A and B2 | Baseline at weeks 4, 8, 12, 14, 16, and 20
Percent Change from Baseline in fasting plasma glucose (FPG) in Cohort A and B2 | Baseline at weeks 4, 8, 12, 14, 16, and 20
Absolute Change from Baseline in fasting plasma glucose in Cohort A and B2 | Baseline, Week 4, 8, 12, 14, 16, and 20 weeks
Percent Change from Baseline in Body Weight in Cohort B1 and B2 | Baseline at weeks 4, 8, 12, 16, and 20
Absolute Change from Baseline in Body Weight in Cohort B1 and B2 | Baseline at weeks 4, 8, 12, 14, 16, and 20

CONTACTS AND LOCATIONS:
Overall Officials: Sin Gon Kim, MD, Principal Investigator — KOREA University Anam Hospital, Seoul, South Korea; Nan Hee Kim, MD, Principal Investigator — KOREA University Asan Hospital in Korea; Soo Lim, MD, Principal Investigator — Seoul National University Bundang Hospital in Korea; Seung-Hwan Lee, MD, Principal Investigator — The Catholic University of KOREA, Seoul St.Mary's Hostital in Korea; Yong-Ho Lee, MD, Principal Investigator — Severance Hostital in Korea; Hyuk-Sang Kwon, MD, Principal Investigator — The Catholic University of KOREA, Yeouido St.Mary's Hostital in Korea; Jang Won Son, MD, Principal Investigator — The Catholic University of KOREA, Bucheon St.Mary's Hostital in Korea; Sang Youl Rhee, MD, Principal Investigator — Kyung Hee University, Medical Center in Korea; In Kyung Jeong, MD, Principal Investigator — Kyung Hee University Hospital at Gangdong in Korea; Jae-Heon Kang, MD, Principal Investigator — Kangbuk Samsung Hospital, Samsung Medical Center in Korea; Jae Hyeon Kim, MD, Principal Investigator — Samsung Medical Center in Korea; Kyung Wan Min, MD, Principal Investigator — Nowon Eul Ji Medical Center, Eul Ji University in Korea; Jun Hwa Hong, MD, Principal Investigator — Daejeon Eul Ji Medical Center, Eul Ji University in Korea; Kyu Chang Won, MD, Principal Investigator — Yeungnam University Medical Center in Korea
Locations (14):
- South Korea (14):
  - The Catholic University of KOREA, Bucheon St.Mary's Hostital, Bucheon-si
  - Yeungnam University Medical Center, Daegu
  - Daejeon Eul Ji Medical Center, Eul Ji University, Daejeon
  - Seoul National University Bundang Hospital, Seongnam
  - Kangbuk Samsung Hospital, Samsung Medical Center, Seoul
  - KOREA University Anam Hospital, Seoul
  - KOREA University Asan Hospital, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul
  - Kyung Hee University, Medical Center, Seoul
  - Nowon Eul Ji Medical Center, Eul Ji University, Seoul
  - Samsung Medical Center, Seoul
  - Severance Hostital, Seoul
  - The Catholic University of KOREA, Seoul St.Mary's Hostital, Seoul
  - The Catholic University of KOREA, Yeouido St.Mary's Hostital in Korea, Seoul